CLINICAL TRIAL: NCT02881177
Title: The Effects of Intranasal Oxytocin on Mixed HIV Sero-status, Methamphetamine-using Men Who Have Sex With Men
Brief Title: Oxytocin HIV Meth Study
Acronym: OHM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Christopher Stauffer, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16-20360
Record Dates: First submitted 2016-08-22; First posted 2016-08-26 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Amphetamine Use Disorders
Keywords: oxytocin; tolerability; HIV; men who have sex with men (MSM); addiction
MeSH Terms: conditions — Homosexuality; Behavior, Addictive | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): Oxytocin 40 International Units (IU) intranasal administration prior to six Motivational Interviewing Group Therapy (MIGT) sessions.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo 40 International Units (IU) intranasal administration prior to six Motivational Interviewing Group Therapy (MIGT) sessions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 40 IU
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — 40 IU
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to determine the tolerability, feasibility, and preliminary effectiveness of intranasal oxytocin administration prior to motivational enhancement group therapy sessions on laboratory-based measures of addiction, social connectedness, and stress responsivity in methamphetamine(meth)-using men who have sex with men (MSM). The investigators propose a randomized, double-blind, study of intranasal oxytocin versus placebo 40 IU prior to each of six Motivational Interviewing Group Therapy (MIGT) sessions in 28 mixed HIV sero-status MSM initiating treatment for amphetamine use disorder.

DETAILED DESCRIPTION:
The high prevalence of amphetamine use disorder (AUD) among men who have sex with men (MSM) leads to significant health disparities, including increased risk for HIV sero-conversion. Reducing methamphetamine use mitigates HIV risk. Currently no psychopharmacological agent exists for the treatment of AUD; innovative interventions are desperately needed. Oxytocin, a social neuropeptide, has well-studied anti-addiction effects in animal models of substance dependence. The use of intranasal oxytocin for a variety of human substance use disorders is under early investigation, although no one has studied oxytocin's effects in AUD. In other populations, oxytocin's effects are known to vary depending on social context. Psychosocial treatment alone has been shown to reduce methamphetamine and HIV risk in MSM at a community-based clinic in San Francisco, The Stonewall Project. The investigators propose a randomized, double-blind pilot study of psychopharmacological-psychosocial combination therapy, administration of intranasal oxytocin versus placebo prior to six Motivational Interviewing Group Therapy (MIGT) sessions, in 28 mixed HIV sero-status MSM initiating treatment for AUD. The investigators aim to assess: 1) tolerability, 2) feasibility for larger randomized controlled trials, and 3) exploratory measures of efficacy, including: a) urine levels of methamphetamine and metabolites, b) methamphetamine craving, c) engagement in MIGT through third-party coding of videotaped group sessions and self-reported measures of group connectedness, d) psychophysiological stress responses to group engagement, and e) sexual risk taking.

ELIGIBILITY:
Inclusion Criteria:

1. One documented urine toxicology screen positive for meth in the past month
2. Considering initiating treatment for Methamphetamine Use Disorder or initiated treatment within the past month
3. History of sexual contact with men.

Exclusion Criteria:

1. Urine toxicology screen positive for heroin in the past month
2. Meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for current psychotic disorder, severe neuropsychological disorder, current moderate-severe alcohol use disorder, or suicidal or homicidal ideation with intent within the past 90-days
3. Hemodialysis or inability to produce urine samples
4. Sensitivity to: E 216, E 218, and chlorobutanol hemihydrate (preservatives used in nasal spray)
5. Nasal Obstruction or discharge
6. Using Hormone supplementation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Side effect profile | 6 weeks
  Aim 1: To examine the tolerability of repeated oxytocin dosing in MSM who use meth.
  Hypothesis 1: There will be no difference in side effect profiles for those receiving oxytocin (40 IU) versus placebo prior to each of six MIGT sessions, and there will be no study-related adverse events.

SECONDARY OUTCOMES:
Recruitment Rates | 6 weeks
  Aim 2: To determine the feasibility of implementing a larger randomized controlled trial of oxytocin dosing in meth-using MSM.
  Hypothesis 2: This community-based pilot study will recruit and enroll 38 individuals within 6 months and have retention rates ≥75%. The investigators will collect effect size data to be used in planning the sample size of larger clinical trials. The investigators will collect pilot validation data for our exploratory measures and paradigms.
urine toxicology | 6 weeks
  Although efficacy is not the primary aim of this pilot study, following administration of 40 IU intranasal oxytocin compared to placebo prior to six MIGT sessions the investigators expect to see trends toward reduction in meth-positive urine toxicology screens.
Meth Craving Questionnaire-Brief (MCQ-Br) | 6 weeks
  Although efficacy is not the primary aim of this pilot study, following administration of 40 IU intranasal oxytocin compared to placebo prior to six MIGT sessions the investigators expect to see trends toward reduced self-reported meth craving as measured by the MCQ-Br.
attendance rate | 6 weeks
  Although efficacy is not the primary aim of this pilot study, following administration of 40 IU intranasal oxytocin compared to placebo prior to six MIGT sessions the investigators expect to see trends toward improved attendance.
Group Questionnaire | 6 weeks
  Although efficacy is not the primary aim of this pilot study, following administration of 40 IU intranasal oxytocin compared to placebo prior to six MIGT sessions the investigators expect to see trends toward increased therapeutic alliance as measured by the Group Questionnaire.
heart rate variability | 6 weeks
  Although efficacy is not the primary aim of this pilot study, following administration of 40 IU intranasal oxytocin compared to placebo prior to six MIGT sessions the investigators expect to see trends toward increased heart rate variability, a marker of parasympathetic control.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Stauffer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thorson KR, McKernan SM, West TV, Woolley JD, Mendes WB, Stauffer CS. Oxytocin increases physiological linkage during group therapy for methamphetamine use disorder: a randomized clinical trial. Sci Rep. 2021 Oct 25;11(1):21004. doi: 10.1038/s41598-021-99957-8. PMID 34697392
- [Derived] Stauffer CS, Moschetto JM, McKernan SM, Hsiang E, Borsari B, Woolley JD. Oxytocin-enhanced motivational interviewing group therapy for methamphetamine use disorder in men who have sex with men: study protocol for a randomized controlled trial. Trials. 2019 Feb 21;20(1):145. doi: 10.1186/s13063-019-3225-7. PMID 30791944